CLINICAL TRIAL: NCT02934724
Title: Impact of HPV Vaccine On The Prevalence Of Human Papillomavirus In Mouth And Vagina In Norway
Brief Title: Impact of HPV Vaccine On The Prevalence Of HPV In Norway
Status: Completed | Type: Observational
Sponsor: Oslo University Hospital (Other)
Collaborators: University Hospital, Akershus (Other)
Responsible Party: Principal Investigator, Espen Enerly, Dr Scient, Oslo University Hospital
Other Study IDs: 2014/2333
Record Dates: First submitted 2016-10-13; First posted 2016-10-17 (Estimated); Last update posted 2020-12-14 (Actual); Status verified 2020-12

CONDITIONS: Cervical Intraepithelial Neoplasia; Cervical Cancer; Oropharyngeal Cancer
Keywords: HPV vaccines; HPV-6; HPV-11; HPV-16; HPV-18; Gardasil
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Neoplasms; Oropharyngeal Neoplasms | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Self samples from vagina and the oral cavity
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Vaccinated: Women born in 1997, resident to Norway in 2009, vaccinated by the quadrivalent HPV vaccine.
  Interventions:
  * Self sample from vagina using Rover's Evalyn Brush
  * Self sample from the oral cavity using COPAN's FloqSwab
  * Questionnaire
  Interventions: Procedure: Self sample from vagina; Procedure: Self sample from the oral cavity; Other: Questionnaire
- Un-vaccinated: Women born in 1997, resident to Norway in 2009, not vaccinated by the quadrivalent HPV vaccine
  Interventions:
  * Self sample from vagina using Rover's Evalyn Brush
  * Self sample from the oral cavity using COPAN's FloqSwab
  * Questionnaire
  Interventions: Procedure: Self sample from vagina; Procedure: Self sample from the oral cavity; Other: Questionnaire

INTERVENTIONS:
Procedure: Self sample from vagina — Self sample using The Rover's Evalyn Brush
Procedure: Self sample from the oral cavity — Self sample using COPAN FloqSwab
Other: Questionnaire — Questionnaire about vaccination status and sexual behaviour

SUMMARY:
The overall aim of the study is to assess the effect of school-based Human Papillomavirus (HPV) vaccination by comparing type-specific HPV prevalence between vaccinated and non-vaccinated women born in 1997. Women born in 1997, residence to Norway in 2009 (the year of vaccine initiation of the 1997-cohort) are invited to participate in the study.

DETAILED DESCRIPTION:
This cohort is amongst the first that was offered HPV vaccine in an organized vaccination programme globally. The women will be recruited through Facebook ads. The study will enable us to measure differences in the prevalence of HPV types in vagina and the mouth between vaccinated and non-vaccinated young women in Norway.

The womens vaccination status will be validated by linkage to the Norwegian Immunisation Registry (SYSVAK) and their residence status will be validated through linkage to the Norwegian Population Registry.

ELIGIBILITY:
Inclusion Criteria:

* Female
* Born in 1997
* Resident of Norway in 2009

Exclusion Criteria:

* Male
* Born before or after 1997
* Non-resident of Norway in 2009

Ages: 18 Years to 20 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Women resident to Norway in 2009
Sampling Method: Non-Probability Sample
Enrollment: 315 (Actual)
Dates: Start 2016-11 (Actual); Primary Completion 2017-02 (Actual); Study Completion 2017-02 (Actual)

PRIMARY OUTCOMES:
Vaginal and oral HPV-6, HPV-11, HPV-16 and HPV-18 prevalence | Within 2 months after self-collection of specimens
  The differences in HPV types prevalence among vaccinees and non-vaccinees. HPV types will be assessed individually and combined.

SECONDARY OUTCOMES:
Description of oral and vaginal overall genotype distribution among vaccinated and non-vaccination participants | Within 2 months after self-collection of specimens

CONTACTS AND LOCATIONS:
Overall Officials: Espen Enerly, Dr Scient, Principal Investigator — Oslo University Hospital; Giske Ursin, Dr.Med, Study Director — Oslo University Hospital
Locations (1):
- Oslo University Hospital, Cancer Registry of Norway, Oslo, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] PLOS ONE Staff. Correction: An observational study comparing HPV prevalence and type distribution between HPV-vaccinated and -unvaccinated girls after introduction of school-based HPV vaccination in Norway. PLoS One. 2019 Dec 12;14(12):e0226706. doi: 10.1371/journal.pone.0226706. eCollection 2019. PMID 31830145
- [Result] Enerly E, Flingtorp R, Christiansen IK, Campbell S, Hansen M, Myklebust TA, Weiderpass E, Nygard M. An observational study comparing HPV prevalence and type distribution between HPV-vaccinated and -unvaccinated girls after introduction of school-based HPV vaccination in Norway. PLoS One. 2019 Oct 10;14(10):e0223612. doi: 10.1371/journal.pone.0223612. eCollection 2019. PMID 31600341